CLINICAL TRIAL: NCT06911268
Title: The Effect of Flipped Learning on Nursing Students' Knowledge and Skills of Inhaler Drug Administration
Brief Title: Flipped Learning on Inhaler Drug Administration
Status: Completed | Type: Observational
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Sponsor
Other Study IDs: Semanur Bilgiç 1(inhaler)
Record Dates: First submitted 2025-02-04; First posted 2025-04-04 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2024-11

CONDITIONS: Nursing Students
Keywords: inhalation drugs; nursing student; flipped learning

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the study, it was aimed to evaluate the effect of inverted classroom teaching method on nursing students' inhaler drug application knowledge and skills.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is an important public health problem characterised by airflow limitation and persistent respiratory symptoms. The World Health Organisation reports that 384 million people worldwide live with COPD and approximately 3 million people die each year due to this disease. Effective management of the disease is of great importance for both individual health and public health. Successful disease management improves the quality of life of patients, slows the progression of the disease, reduces the frequency of attacks, and prevents morbidity and mortality. For this purpose, treatment management is recognised as a building block.

Various drugs such as bronchodilators, anti-inflammatory drugs and mucolytics are used in the treatment of COPD. These drugs are usually given in inhaler form and each inhaler drug is administered with a different technique. These techniques include metered dose inhalers, dry powder inhalers (aeroliser, breezhaler, discus, easyhaler, ellipta, handihaler, sonohaler), soft mist inhalers (vapour aerosols) and nebulisers. However, all these drugs can be effective only when applied with the correct technique. Improper use of inhalers decreases patient compliance, increases the number and frequency of attacks, and may cause the dose to be increased by the physician. For this purpose, patient education about inhaler devices is very important. Based on this, nurses should know, apply and teach the correct inhaler techniques to patients.

Nurses learn theoretical and psychomotor skills, especially inhaler drug applications, during the education process. An effective and successful education both increases the knowledge of nurses and improves their psychomotor skills for practice. In this context, the application of different teaching methods in the learning of complex information and the application of skills provides comprehensibility and retention. These methods are of great importance in critical thinking ability, clinical performance, knowledge competence and transformation of knowledge into clinical skills.

One of these methods, the flipped classroom model, is based on the principle of integrating the activities carried out in the classroom outside the classroom and the teaching activities carried out outside the classroom inside the classroom. In the literature, it is emphasised that nursing students should know the correct use of inhalers and should be skilled. However, studies on this subject are quite limited and it is recommended that more studies be conducted on this subject.

ELIGIBILITY:
Inclusion Criteria:

* Students who were attending the course on the date the research data were collected,
* who had not received training on respiratory system diseases and inhaler drug applications before,
* who had a phone or computer with internet access and who agreed to participate in the research

Exclusion Criteria:

* Students who are absent from the course and
* do not participate in one of the pre-test, post-test and follow-up test

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: nursing student
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
Knowledge test scoring to measure students' knowledge levels | 7 weeks
  nursing students' level of knowledge and skills of Inhaler drug administration

CONTACTS AND LOCATIONS:
Locations (1):
- Bilecik Şeyh Edebali University, Bilecik, Bilecik, Turkey (Türkiye)